CLINICAL TRIAL: NCT00454571
Title: A Randomized, Phase II Study of GW786034 (Pazopanib) in Stage D0 Relapsed Androgen Sensitive Prostate Cancer Following Limited GnRH Agonist Therapy
Brief Title: Pazopanib Hydrochloride After Leuprolide Acetate or Goserelin Acetate in Treating Patients With Relapsed Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00202; N01CM62201 (NIH); CDR0000538086 (Registry Identifier: PDQ (Physician Data Query)); 14954A
Record Dates: First submitted 2007-03-27; First posted 2007-03-30 (Estimated); Results first posted 2016-02-10 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2012-09

CONDITIONS: Recurrent Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — pazopanib; Leuprolide; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pazopanib (Experimental): Patients receive pazopanib hydrochloride PO QD on days 1-28 after treatment with leuprolide acetate and goserelin acetate. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: pazopanib hydrochloride; Drug: leuprolide acetate; Drug: goserelin acetate
- Observation (Active Comparator): Patients undergo observation after treatment with leuprolide acetate and goserelin acetate.
  Interventions: Drug: leuprolide acetate; Drug: goserelin acetate

INTERVENTIONS:
Drug: pazopanib hydrochloride — Given PO
  Other Names: GW786034B; Votrient
  Arms: Pazopanib
Drug: leuprolide acetate
  Other Names: Enantone; LEUP; Lupron; Lupron Depot
Drug: goserelin acetate
  Other Names: ICI-118630; ZDX; Zoladex

SUMMARY:
This randomized phase II trial is studying how well pazopanib hydrochloride works after leuprolide or goserelin in treating patients with relapsed prostate cancer. Pazopanib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Androgens can cause the growth of prostate cancer cells. Antihormone therapy, such as leuprolide acetate or goserelin acetate, may lessen the amount of androgens made by the body. Giving pazopanib after leuprolide or goserelin may be an effective treatment for prostate cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine if pazopanib hydrochloride is able to increase time to progression, as measured by prostate-specific antigen (PSA), after 6 months of limited gonadotropin-releasing hormone (GnRH) agonist therapy comprising leuprolide acetate or goserelin in patients with androgen-sensitive relapsed stage D0 prostate cancer.

SECONDARY OBJECTIVES:

I. Determine the adverse events in patients treated with this regimen. II. To monitor for changes in testosterone in relationship to pazopanib therapy versus observation.

OUTLINE:

Patients receive androgen blockade comprising GnRH agonist therapy (e.g., leuprolide acetate or goserelin acetate) for 6 months. Patients who develop metastases or have PSA progression while on GnRH agonist therapy are removed from the study and placed on total androgen blockade. The remaining patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive pazopanib hydrochloride orally (PO) once daily (QD) on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients undergo observation.

After completion of study treatment, patients are followed up periodically for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed prostate cancer

  * Stage D0
* Must have undergone some definitive local therapy for prostate cancer
* Must be free of macrometastatic disease, as evidenced by computed tomography (CT) scan and bone scan, if serum PSA ≥ 10 ng/mL prior to GnRH agonist therapy
* Progressive disease meeting the following criteria: NOTE: Patients who have undergone a prostatectomy and have two detectable, rising serum PSA levels are eligible

  * Two consecutive rises in PSA above nadir recorded after definite local therapy
  * Serum PSA concentrations must have absolute value of > 0.5 ng/mL (separated by ≥ 2 weeks) prior to beginning GnRH agonist therapy
* PSA < 0.5 ng/mL
* Testosterone < 30 ng/mL
* No measurable disease
* No brain metastases requiring steroid or anticonvulsant therapy
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2 OR Karnofsky PS 60- 100%
* Prothrombin time (PT)/international normalization ratio (INR)/partial thromboplastin time (PTT) ≤ 1.2 times upper limit of normal (ULN)
* Bilirubin normal
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN OR creatinine clearance > 50 mL/min
* Proteinuria ≤ 1+ on 2 consecutive dipsticks > 1 week apart
* Urine protein: creatinine ratio < 1 OR urine protein < 1.0 g/24 hours
* Fertile patients must use effective double-barrier contraception during study therapy OR completely abstain from sexual intercourse 14 days prior to, during, and for ≥ 21 days after completion of study therapy
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to pazopanib hydrochloride or to other agents used in the study
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Psychiatric illness or social situations that would preclude compliance with study requirements
* No human immunodeficiency virus (HIV) positivity
* No condition that impairs the ability to swallow and retain pazopanib hydrochloride tablets, including any of the following:

  * Gastrointestinal tract disease resulting in an inability to take oral medication
  * Requirement for intravenous (IV) alimentation
  * Prior surgical procedures affecting absorption
  * Active peptic ulcer disease
* No other conditions, including any of the following:

  * Serious or nonhealing wound, ulcer, or bone fracture
  * Abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
  * Cerebrovascular accident within the past 6 months
  * Myocardial infarction, admission for unstable angina, cardiac angioplasty, or stenting within the past 6 months
  * Venous thrombosis within the past 12 weeks
  * New York Heart Association (NYHA) class III or IV heart failure

    * History of currently treated asymptomatic NYHA class II heart failure allowed
* Systolic blood pressure (BP) ≤ 140 mm Hg and diastolic BP ≤ 90 mm Hg

  * Prior initiation or adjustment of BP medication allowed provided that the average of 3 BP readings at a visit prior to enrollment is < 140/90 mm Hg
* More than 3 months since prior antiandrogen
* More than 4 months since prior orchiectomy or implantable luteinizing LHRH agonist
* No prior GnRH agonists except for neoadjuvant or adjuvant therapy associated with local therapy

  * Patients who have started a GnRH agonist for micrometastatic disease after local therapy allowed provided the following criteria are met:

    * Progressive disease
    * Willing to discontinue therapy before 6 months have elapsed
    * Have signed consent prior to completing 6 months of the initial hormone therapy
    * Are within 4 months of initiating GnRH agonist therapy
* No prior or concurrent GnRH antagonist therapy
* No concurrent ketoconazole
* No concurrent cytochrome P450 2C9 (CYP2C9) substrates, including any of the following:

  * Anticoagulants (e.g., warfarin [therapeutic doses only])

    * Low molecular weight heparin or prophylactic low-dose warfarin allowed
  * Oral hypoglycemics (e.g., glipizide, glyburide, tolbutamide, glimepiride, or nateglinide)
  * Ergot derivatives (e.g., dihydroergotamine, ergonovine, ergotamine, or methylergonovine)
  * Neuroleptics (e.g., pimozide)
  * Erectile dysfunction agents (e.g., sildenafil, tadalafil, or vardenafil)
  * Antiarrhythmics (e.g., bepridil, flecainide, lidocaine, mexiletin, amiodarone, quinidine, or propafenone)
  * Immune modulators (e.g., cyclosporine, tacrolimus, or sirolimus)
  * Miscellaneous medications (e.g., theophylline, quetiapine, risperidone, tacrine, clozapine, or atomoxetine)
* No concurrent medications associated with the risk of QTc prolongation and/or Torsades de Pointes

  * Replacement of drugs that do not carry these risks allowed
* No other concurrent non-Food and Drug Administration (FDA)-approved agents

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Posadas, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

REFERENCES:
- [Result] Ward JE, Karrison T, Chatta G, Hussain M, Shevrin D, Szmulewitz RZ, O'Donnell PH, Stadler WM, Posadas EM. A randomized, phase II study of pazopanib in castrate-sensitive prostate cancer: a University of Chicago Phase II Consortium/Department of Defense Prostate Cancer Clinical Trials Consortium study. Prostate Cancer Prostatic Dis. 2012 Mar;15(1):87-92. doi: 10.1038/pcan.2011.49. Epub 2011 Oct 18. PMID 22006050

RESULTS

PARTICIPANT FLOW:
Groups:
- Pazopanib, Leuprolide Acetate, and Goserelin Acetate: Patients receive pazopanib hydrochloride PO QD on days 1-28 after treatment with leuprolide acetate and goserelin acetate. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  pazopanib hydrochloride: Given PO
  leuprolide acetate
  goserelin acetate
- Leuprolide Acetate and Goserelin Acetate Only: Patients undergo observation after treatment with leuprolide acetate and goserelin acetate.
  leuprolide acetate
  goserelin acetate
Period: Overall Study
Arm/Group | Pazopanib, Leuprolide Acetate, and Goserelin Acetate | Leuprolide Acetate and Goserelin Acetate Only
Started | 18 | 19
Completed | 5 | 13
Not Completed | 13 | 6
Not completed — Adverse Event | 2 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 10 | 5

BASELINE CHARACTERISTICS:
Population: Baseline demographics data for this multi-center trial are only available for participants at The University of Chicago with known study arm assignment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pazopanib, Leuprolide Acetate, and Goserelin Acetate | Leuprolide Acetate and Goserelin Acetate Only | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Continuous [Median (Full Range); unit: years] | 74 [60 to 90] | 71 [63 to 83] | 72 [60 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 18 | 19 | 37

OUTCOME MEASURES:

1. Primary Outcome: Median Time to PSA Progression
Description: The median time to disease progression for the therapy and observation groups will be estimated using the Kaplan-Meier estimate and compared using the log-rank test.
Time Frame: Baseline, every 4 weeks during treatment, and up to 12 months after completion of study treatment
Population: Patients were taken off study early, so many survival times were censored. At no point during the study did the proportion of subjects who progressed drop to 50%. Thus, it was not possible to calculate median time to disease progression.
Arm/Group | Pazopanib, Leuprolide Acetate, and Goserelin Acetate | Leuprolide Acetate and Goserelin Acetate Only
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Median PSA Progression-free Survival
Description: Kaplan-Meier estimates for PSA progression-free survival will be computed for the pazopanib and active surveillance groups and compared using the log rank test. The outcome measure is median PSA progression-free survival time.
Time Frame: Time from randomization to PSA progression or death from any cause
Population: Patients were taken off study early, so many survival times were censored. At no point during the study did the proportion of subjects who progressed drop to 50%. Thus, it was not possible to calculate median time to PSA progression.
Arm/Group | Pazopanib, Leuprolide Acetate, and Goserelin Acetate | Leuprolide Acetate and Goserelin Acetate Only
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Pazopanib, Leuprolide Acetate, and Goserelin Acetate | Leuprolide Acetate and Goserelin Acetate Only
Serious Adverse Events (participants affected / at risk) | 5/18 | 0/19
Other Adverse Events (participants affected / at risk) | 16/18 | 2/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib, Leuprolide Acetate, and Goserelin Acetate (N=18) | Leuprolide Acetate and Goserelin Acetate Only (N=19)
Alanine aminotransferase increased (Investigations) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib, Leuprolide Acetate, and Goserelin Acetate (N=18) | Leuprolide Acetate and Goserelin Acetate Only (N=19)
Anemia (Blood and lymphatic system disorders) | 4 | 0 — A disorder characterized by an reduction in the amount of hemoglobin in 100 ml of blood.
Tinnitus (Ear and labyrinth disorders) | 1 | 0 — A disorder characterized by noise in the ears, such as ringing, buzzing, roaring or clicking.
Blurred vision (Eye disorders) | 1 | 0 — A disorder characterized by visual perception of unclear or fuzzy images.
Eye disorders - Other (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 — A disorder characterized by a sensation of marked discomfort in the abdominal region.
Constipation (Gastrointestinal disorders) | 2 | 1 — A disorder characterized by irregular and infrequent or difficult evacuation of the bowels.
Diarrhea (Gastrointestinal disorders) | 12 | 0 — A disorder characterized by frequent and watery bowel movements.
Dyspepsia (Gastrointestinal disorders) | 3 | 0 — A disorder characterized by an uncomfortable, often painful feeling in the stomach, resulting from impaired digestion. Symptoms include burning stomach, bloating, heartburn, nausea and vomiting.
Esophagitis (Gastrointestinal disorders) | 1 | 0 — A disorder characterized by inflammation of the esophageal wall.
Flatulence (Gastrointestinal disorders) | 2 | 0 — A disorder characterized by a state of excessive gas in the alimentary canal.
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0 — A disorder characterized by the presence of dilated veins in the rectum and surrounding area.
Mucositis oral (Gastrointestinal disorders) | 1 | 0 — A disorder characterized by inflammation of the oral mucosal.
Nausea (Gastrointestinal disorders) | 3 | 0 — A disorder characterized by a queasy sensation and/or the urge to vomit.
Oral pain (Gastrointestinal disorders) | 1 | 0 — A disorder characterized by a sensation of marked discomfort in the mouth, tongue or lips.
Stomach pain (Gastrointestinal disorders) | 1 | 0 — A disorder characterized by a sensation of marked discomfort in the stomach.
Vomiting (Gastrointestinal disorders) | 1 | 0 — A disorder characterized by the reflexive act of ejecting the contents of the stomach through the mouth.
Edema face (General disorders) | 1 | 0 — A disorder characterized by swelling due to excessive fluid accumulation in facial tissues.
Fatigue (General disorders) | 9 | 0 — A disorder characterized by a state of generalized weakness with a pronounced inability to summon sufficient energy to accomplish daily activities.
Pain (General disorders) | 3 | 1 — A disorder characterized by the sensation of marked discomfort, distress or agony.
Alanine aminotransferase increased (Investigations) | 7 | 0 — A finding based on laboratory test results that indicate an increase in the level of alanine aminotransferase (ALT or SGPT) in the blood specimen.
Alkaline phosphatase increased (Investigations) | 1 | 0 — A finding based on laboratory test results that indicate an increase in the level of alkaline phosphatase in a blood specimen.
Aspartate aminotransferase increased (Investigations) | 8 | 0 — A finding based on laboratory test results that indicate an increase in the level of aspartate aminotransferase (AST or SGOT) in a blood specimen.
Blood bilirubin increased (Investigations) | 1 | 0 — A finding based on laboratory test results that indicate an abnormally high level of bilirubin in the blood. Excess bilirubin is associated with jaundice.
Creatinine increased (Investigations) | 1 | 0 — A finding based on laboratory test results that indicate increased levels of creatinine in a biological specimen.
Lymphocyte count decreased (Investigations) | 2 | 0 — A finding based on laboratory test results that indicate a decrease in number of lymphocytes in a blood specimen.
Platelet count decreased (Investigations) | 3 | 0 — A finding based on laboratory test results that indicate a decrease in number of platelets in a blood specimen.
Weight gain (Investigations) | 0 | 1 — A finding characterized by an increase in overall body weight; for pediatrics, greater than the baseline growth curve.
Weight loss (Investigations) | 3 | 0 — A finding characterized by a decrease in overall body weight; for pediatrics, less than the baseline growth curve.
White blood cell decreased (Investigations) | 2 | 0 — A finding based on laboratory test results that indicate an decrease in number of white blood cells in a blood specimen.
Anorexia (Metabolism and nutrition disorders) | 4 | 0 — A disorder characterized by a loss of appetite.
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 0 — A disorder characterized by laboratory test results that indicate an elevation in the concentration of blood sugar. It is usually an indication of diabetes mellitus or glucose intolerance.
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 — A disorder characterized by laboratory test results that indicate an elevation in the concentration of potassium in the blood; associated with kidney failure or sometimes with the use of diuretic drugs.
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 0 — A disorder characterized by laboratory test results that indicate a low concentration of albumin in the blood.
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 — A disorder characterized by laboratory test results that indicate a low concentration of glucose in the blood.
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0 — A disorder characterized by laboratory test results that indicate a low concentration of magnesium in the blood.
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0 — A disorder characterized by laboratory test results that indicate a low concentration of sodium in the blood.
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 0 — A disorder characterized by laboratory test results that indicate a low concentration of phosphates in the blood.
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 — A disorder characterized by a sensation of marked discomfort in a joint.
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 — A disorder characterized by marked discomfort sensation in the back region.
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0 — A disorder characterized by marked discomfort sensation in the chest wall region.
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 — A disorder characterized by a disturbing sensation of lightheadedness, unsteadiness, giddiness, spinning or rocking.
Dysgeusia (Nervous system disorders) | 3 | 0 — A disorder characterized by abnormal sensual experience with the taste of foodstuffs; it can be related to a decrease in the sense of smell.
Headache (Nervous system disorders) | 4 | 0 — A disorder characterized by a sensation of marked discomfort in various parts of the head, not confined to the area of distribution of any nerve.
Memory impairment (Nervous system disorders) | 1 | 0 — A disorder characterized by a deterioration in memory function.
Nervous system disorders - Other (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 — A disorder characterized by inflammation or degeneration of the peripheral sensory nerves.
Anxiety (Psychiatric disorders) | 1 | 0 — A disorder characterized by apprehension of danger and dread accompanied by restlessness, tension, tachycardia, and dyspnea unattached to a clearly identifiable stimulus.
Libido decreased (Psychiatric disorders) | 0 | 1 — A disorder characterized by a decrease in sexual desire.
Proteinuria (Renal and urinary disorders) | 1 | 0 — A disorder characterized by laboratory test results that indicate the presence of excessive protein in the urine. It is predominantly albumin, but also globulin.
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 | 0
Urinary frequency (Renal and urinary disorders) | 2 | 0 — A disorder characterized by urination at short intervals.
Urinary incontinence (Renal and urinary disorders) | 2 | 1 — A disorder characterized by inability to control the flow of urine from the bladder.
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — A disorder characterized by an inflammation of the nasal mucous membranes caused by an IgE-mediated response to external allergens.
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — A disorder characterized by sudden, often repetitive, spasmodic contraction of the thoracic cavity, resulting in violent release of air from the lungs and usually accompanied by a distinctive sound.
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 0 — A disorder characterized by an uncomfortable sensation of difficulty breathing.
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 0 — A disorder characterized by a decrease in density of hair compared to normal for a given individual at a given age and body location.
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 | 0 — A disorder characterized by an increase in sensitivity of the skin to light.
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 — A disorder characterized by an intense itching sensation.
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 3 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 — A disorder characterized by circumscribed, inflammatory and necrotic erosive lesion on the skin.
Hot flashes (Vascular disorders) | 3 | 1 — A disorder characterized by an uncomfortable and temporary sensation of intense body warmth, flushing, sometimes accompanied by sweating upon cooling.
Hypertension (Vascular disorders) | 9 | 0 — A disorder characterized by a pathological increase in blood pressure; a repeatedly elevation in the blood pressure exceeding 140 over 90 mm Hg.
Hypotension (Vascular disorders) | 1 | 0 — A disorder characterized by a blood pressure that is below the normal expected for an individual in a given environment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less